CLINICAL TRIAL: NCT01015976
Title: A Preliminary Comparison of the Blood Levels of Medications in Obese Subjects Compared to Post-Gastric Bypass Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Collaborators: University of North Dakota (Other)
Responsible Party: Principal Investigator, James Roerig, James L. Roerig, Pharm.D., BCPP, University of North Dakota Department of Clinical Neuroscience, Grand Forks, ND and the Neuropsychiatric Research Institute, Fargo, ND., Neuropsychiatric Research Institute, Fargo, North Dakota
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200803-272
Record Dates: First submitted 2009-10-01; First posted 2009-11-18 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-02

CONDITIONS: Obesity
Keywords: Gastric Bypass; Sertraline; Pharmacokinetics
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post bariatric surgery (Experimental): Roux en Y bariatric surgery
  Interventions: Procedure: bariatric surgery
- Control (Other): No surgery
  Interventions: Other: control

INTERVENTIONS:
Procedure: bariatric surgery — Roux en Y bariatric surgery
  Arms: Post bariatric surgery
Other: control — No surgery
  Arms: Control

SUMMARY:
The purpose of this study is to determine the difference, if any, in the area under the sertraline plasma level time curve (AUC) between patients who are nine to fifteen months post Roux-en-Y Bariatric Surgery and control subjects matched for body mass index (BMI), age and gender.

DETAILED DESCRIPTION:
Secondary objectives include the determination of changes in mean CPmax, Time to CPmax and Volume of Distribution between the two groups. Also, assessment of subject tolerance of sertraline utilizing the UKU side effect rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 60 years.
* Subjects must be of good general health by history and physical exam.
* Five subjects 9 to 15 months past bariatric surgery (Roux-en-Y procedure), no BMI requirement.
* Five subjects matched for body mass index, age and sex to the post bariatric surgery group.
* No contraindications to receiving a single dose of 100 mg of sertraline.
* Women of child bearing potential must be practicing an accepted method of birth control (barrier method or oral contraception) and have a negative pregnancy test at baseline.

Exclusion Criteria:

* Allergy to sertraline or any of its constituents.
* Candidates currently receiving sertraline or any other antidepressant.
* Candidates currently receiving a medication that interacts with sertraline (Zoloft)
* Candidates who are poor metabolizers for the CYP2D6 and/or 2C19 enzymes.
* Candidates experiencing clinically significant, unstable neurological, hepatic, renal or cardiovascular disease.
* Candidates currently or with a past history of meeting DSM-IV diagnostic criteria for schizophrenia, schizoaffective disorder, bipolar disorder.
* Candidates who have participated in an investigational drug study in past 30 days.
* Candidates who meet DSM-IV diagnostic criteria for drug/alcohol abuse or dependency or who have a history of drug/alcohol abuse or dependency.
* Candidates who are pregnant or nursing at time of study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Roerig, PharmD, BCPP, Principal Investigator — Neuropsychiatric Research Institute and University of North Dakota
Locations (1):
- Neuropsychiatric Research Institute, Fargo, North Dakota, United States

REFERENCES:
- See also: Neuropsychiatric Research Institute — http://www.nrifargo.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Post surgery group Sertraline : Single dose of 100mg sertraline
- Control Group: active drug
  No surgery matched subjects
Period: Overall Study
Arm/Group | Experimental | Control Group
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Drug: Single arm study, all receive active drug
  Sertraline : Single dose of 100mg sertraline
Arm/Group | Active Drug
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: AUC Post Surgery (n =5) Compared to AUC Control (n=5)
Description: AUC of surgery group compared to the AUC of control group
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 3.5, 4.5, 6.5, 8.5, 10.5 hours
Population: Per protocol
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Groups:
- Control: Single arm study, all receive active drug
  Sertraline : Single dose of 100mg sertraline
Arm/Group | Control
Number analyzed (Participants) | 10
ng-hr/mL
  Post surgery | 124.4 (55.5)
  Control | 314.8 (129.6)

ADVERSE EVENTS:
Groups:
- Active Drug: Two arm study, all receive active drug
  Sertraline : Single dose of 100mg sertraline
Arm/Group | Active Drug
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
small sample size absence of men in either group. short data collection period, characterization of the linear elimination phase of the AUC was not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No